CLINICAL TRIAL: NCT06698315
Title: Tailored Interventions for Patient Safety: an Evidence-based Approach to Reduce Falls in Adult Patients
Brief Title: Evidence-based Approach to Reduce Falls in Adult Patients
Status: Recruiting | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 011.NUR.2024.R
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Falls with Injuries
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observation — Medical Records Chart Review

SUMMARY:
The project aims to promote patient safety and quality care by reducing preventable falls and falls with injuries using an evidence-based solution.

DETAILED DESCRIPTION:
The project aims to promote patient safety and quality care by reducing preventable falls and falls with injuries using an evidence-based solution: the Fall Tailoring Interventions for Patient Safety (TIPS) intervention. The three objectives include: (a) developing personalized fall prevention interventions for high-risk patients, (b) engaging patients and families in fall prevention initiatives, and (c) promoting effective communication among teams using a bedside visual tool.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) inpatients admitted for various medical-surgical conditions in 3 Medical unit at MRMC. All patients will be included in the project except those diagnosed with psychiatric conditions and cognitive impairments.

Exclusion Criteria:

* Patients with psychiatric conditions and cognitive impairments will be excluded from the project. This assessment is routine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with psychiatric conditions and cognitive impairments will be excluded from the project. This assessment is routine.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Determine if the Fall TIPS initiative is effective at reducing falls at MRMC. | through study completion, up to 18 months
  Data will be collected from Verge and EPIC reports. To ensure intervention effectiveness, monitoring will be done through chart audits and staff reporting. EPIC slicer dicer generates customized reports, enhancing EHR effectiveness (Ayaad et al., 2022).

CONTACTS AND LOCATIONS:
Overall Officials: ELIZABETH D AARON, MSN, Principal Investigator — METHODIST RICHARDSON MEDICAL CENTER
Locations (1):
- Methodist Dallas Medical Center- Clinical Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No